CLINICAL TRIAL: NCT03199898
Title: Reliability Testing of Silverman-Andersen Retraction Score in Preterm Infants
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/588
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2019-07

CONDITIONS: Premature Birth
Keywords: Lung/Growth & Development; Respiration, artificial; Reproducibility of Results; Observer Variation
MeSH Terms: conditions — Premature Birth; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 34-32 GA: premature infants born <34,6-32,1 weeks of gestational age (GA) receiving different types of non-invasive and invasive respiratory support, and severity of respiratory distress assessed by Silverman-Andersen Retraction Score.
  Interventions: Diagnostic Test: Silverman-Andersen Retraction Score
- 32-28 GA: premature infants born <32-28,1 weeks of gestational age (GA) receiving different types of non-invasive and invasive respiratory support, and severity of respiratory distress assessed by Silverman-Andersen Retraction Score.
  Interventions: Diagnostic Test: Silverman-Andersen Retraction Score
- 28-23 GA: premature infants born <28-23,0 weeks of gestational age (GA) receiving different types of non-invasive and invasive respiratory support, and severity of respiratory distress assessed by Silverman-Andersen Retraction Score.
  Interventions: Diagnostic Test: Silverman-Andersen Retraction Score

INTERVENTIONS:
Diagnostic Test: Silverman-Andersen Retraction Score — The Silverman-Andersen Retraction Score (SAs) is used to assess severity of respiratory distress in newborn and preterm infants without respiratory support.The score comprises 4 inspiratory categories of movements (thoraco-abdominal, intercostal, xiphoid, and chin movements) and one expiratory category (grunting).
  Other Names: SAs

SUMMARY:
Depending on their gestational age, preterm infants need several weeks with different types of breathing-support due to immature development of the lungs, respiratory muscles, chest-wall and respiratory center in the brain. WHO's recommendation on interventions to improve preterm birth outcomes underline the need for more research on respiratory support in infants born preterm. This study will test inter-rater and intra-rater reliability of the Silverman-Andersen Retraction Score, which is a systematic clinical scoring tool for the respiratory work and the severity of respiratory distress in preterm infants. It will examine if there is consistency in the assessments done by doctors and nurses, and also if the observations correlate with technological monitoring. This easy to use scoring tool will help to determine the grade of respiratory distress, to assess respiratory exacerbation, to decide when to start weaning from respiratory support, and to give the best respiratory treatment to the child. This study will contribute to optimize care for preterm infants with respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* born <35 weeks gestational age

Exclusion Criteria:

* need of muscle relaxation
* hemodynamic instability

Ages: 2 Weeks to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants born <35 weeks of gestational age. the included infants will be stratified in 3 gestational age groups.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
inter-rater reliability of Silverman-Andersen Retraction Score | 2 weeks
  observers will be pediatric physicians and nurses experienced in the newborn intensive care unit (NICU)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Selvaag, md, Study Director — St. Olavs Hospital
Locations (2):
- Norway (2):
  - Levanger Hospital, Levanger
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brenne H, Follestad T, Bergseng H, Eriksen BH, Soraunet K, Grunewaldt KH. Inter-rater reliability of the Silverman and Andersen index-a measure of respiratory distress in preterm infants. PLoS One. 2023 Jun 30;18(6):e0286655. doi: 10.1371/journal.pone.0286655. eCollection 2023. PMID 37390074